CLINICAL TRIAL: NCT05517278
Title: Clinical Evaluation of the Next Science SurgX Antimicrobial Wound Gel Impact on Surgical Site Complications
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding no longer available
Sponsor: Northwell Health (Other)
Collaborators: Next Science TM (Industry)
Responsible Party: Principal Investigator, Giles Scuderi, Orthopaedic Surgery, Joint Reconstruction, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1050
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Total Hip Arthroplasty; Total Knee Arthroplasty
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): The treatment group will receive SurgX™ Antimicrobial Wound Gel™ applied over incision after closure and then re-applied at first dressing change on day of discharge in addition to standard of care.
  Interventions: Other: SurgX Antimicrobial Wound Gel
- Control Group (Other): The control group will receive standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: SurgX Antimicrobial Wound Gel — In addition to standard of care, at time of surgery, SurgX applied on the incision after closure and then re-applied at the time of first bandage change on day of discharge.
  Arms: Treatment Group
Other: Standard of Care — The control group will receive standard of care.
  Arms: Control Group

SUMMARY:
This is a single-site, prospective, clinical study of subjects that are scheduled to undergo either total hip or total knee arthroplasties. It is anticipated that surgical wounds treated with SurgX will exhibit reduced surgical site complication rates and improved post-operative treatment outcomes by potentially decreasing site bioburden of both free-floating and biofilm-entrenched organisms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years or older
2. Scheduled to undergo primary hip or knee arthroplasty
3. Willing and able to comply with all study procedures and be available for the duration of the study
4. Provide signed and dated informed consent

Exclusion Criteria:

1. Unable to provide signed and dated informed consent
2. Unable or unwilling to comply with all study-related procedures
3. Known history of allergic reaction to any of the study products or its components, including any products used for standard of care (such as dressings or any coverings)
4. Subject with any mental impairment or condition that would make them unable to properly consent without use of LAR or additional subject protections
5. Subjects from a vulnerable population, in accordance with 45 CFR 46 Subparts B, C, and D

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Surgical site complication | within 12 weeks of the index procedure
  Presence/absence of a surgical site complication. Surgical site complications to be defined as meeting at least one of the below criteria:
  1. Bacterial or fungal infection as confirmed by PCR swabs
  2. Hypertrophic scar formation as diagnosed by in-person assessment via the study investigator
  3. Superficial granuloma formation as diagnosed by in-person assessment via study investigator
  4. Wound dehiscence as diagnosed by in-person assessment via study investigator
  5. Presence of discharge as diagnosed by in-person assessment via study investigator
  6. Presence of wound redness as diagnosed by in-person assessment via study investigator
  7. Presence of stitch abscess as diagnosed by in-person assessment via study investigator
  8. Superficial surgical site infection as diagnosed by in-person assessment via study investigator in accordance with the NHSN SSI Checklist

SECONDARY OUTCOMES:
Wound images | 12 weeks after index procedure
  Third party assessment of wound images taken with Tissue Analytics via blinded assessor to corroborate the investigator's assessment using the below criteria:
  1. Hypertrophic scar formation
  2. Superficial granulation
  3. Wound dehiscence
  4. Discharge
  5. Wound redness
  6. Stitch abscess

CONTACTS AND LOCATIONS:
Overall Officials: Giles Scuderi, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gronbeck C, Cote MP, Lieberman JR, Halawi MJ. Risk stratification in primary total joint arthroplasty: the current state of knowledge. Arthroplast Today. 2019 Feb 5;5(1):126-131. doi: 10.1016/j.artd.2018.10.002. eCollection 2019 Mar. PMID 31020036
- [Background] Doyle DJ, Goyal A, Bansal P, et al. American Society of Anesthesiologists Classification. [Updated 2020 Jul 4]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK441940/
- [Background] Moonesinghe SR, Mythen MG, Das P, Rowan KM, Grocott MP. Risk stratification tools for predicting morbidity and mortality in adult patients undergoing major surgery: qualitative systematic review. Anesthesiology. 2013 Oct;119(4):959-81. doi: 10.1097/ALN.0b013e3182a4e94d. PMID 24195875
- [Background] Bilimoria KY, Liu Y, Paruch JL, Zhou L, Kmiecik TE, Ko CY, Cohen ME. Development and evaluation of the universal ACS NSQIP surgical risk calculator: a decision aid and informed consent tool for patients and surgeons. J Am Coll Surg. 2013 Nov;217(5):833-42.e1-3. doi: 10.1016/j.jamcollsurg.2013.07.385. Epub 2013 Sep 18. PMID 24055383